CLINICAL TRIAL: NCT04416737
Title: Evaluating the Benefits of Physiologic Insulin Delivery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rayhan A. Lal, Med+Peds Endocrinologist, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-57032; 1K23DK122017 (NIH)
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will each come in for 3 visits separated by at least 1 week. During the first two visits they will be randomized to either upper or lower peritoneal injection followed by the other site. During the third visit a subcutaneous injection will be performed to provide comparative data to the standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Upper Peritoneal, then Lower Peritoneal, then Subcutaneous (Experimental): Ultra-fast acting insulin will be injected into the upper peritoneum then lower peritoneum then subcutaneous space.
  Interventions: Drug: Ultra-rapid insulin
- Lower Peritoneal, then Upper Peritoneal, then Subcutaneous (Experimental): Ultra-fast acting insulin will be injected into the lower peritoneum then upper peritoneum then subcutaneous space.
  Interventions: Drug: Ultra-rapid insulin

INTERVENTIONS:
Drug: Ultra-rapid insulin — Following 0.5-3 hours of insulin suspension from insulin pump, participants will receive insulin injection in respective locations (separated by at least 1 week) and then have serial lab measurements (YSI glucose, insulin and glucagon) taken during induced hypoglycemia.

SUMMARY:
In normal physiology insulin is secreted by beta cells into the portal vein. There have been a number of purported benefits among long-term intraperitoneal insulin users. In the present study we will inject ultra-rapid acting insulin into the upper and lower peritoneum under ultrasound guidance and compare it to subcutaneous injection. We will measure glucose, insulin and glucagon following these injections, to assess for benefits in counter-regulatory hormone production and insulin pharmacokinetics.

DETAILED DESCRIPTION:
The eventual goal of this line of work is an implanted insulin pump that delivers insulin automatically into the peritoneum based on continuous glucose data. All prior intraperitoneal pharmacokinetic studies used only concentrated regular insulin, which may be too slow to provide full closed-loop insulin delivery without meal announcement. A description of intraperitoneal ultra-rapid insulin kinetics, as well as counter-regulatory hormonal factors that may counter hypoglycemia is needed. Upper versus lower peritoneal delivery may also affect insulin kinetics. A possible benefit of intraperitoneal insulin is restoration of glucagon response in longstanding diabetes and clearance of insulin by the liver, both of which could provide hypoglycemic rescue in automated insulin delivery systems.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years of age
2. Clinical diagnosis of type 1 diabetes
3. On insulin pump therapy and continuous glucose monitor (CGM) for at least 3 months
4. Ability to safely receive intraperitoneal injection
5. For females, not currently known to be pregnant
6. Understanding and willingness to follow the protocol and sign informed consent
7. Ability to speak, read and write in the language of the investigators

Exclusion Criteria:

1. Diabetic ketoacidosis in the past 3 months
2. Severe hypoglycemia resulting in seizure or loss of consciousness within 3 months prior to enrollment
3. Pregnant or lactating
4. Active infection
5. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol
6. Known cardiovascular events in the last 6 months
7. Known seizure disorder
8. Inpatient psychiatric treatment in the past 6 months
9. Lack of stability on medication 1 month prior to enrollment including antihypertensive, thyroid, anti-depressant or lipid lowering medication.
10. Suspected drug or alcohol abuse
11. Chronic kidney disease (GFR < 60 mL/min/1.73m^2)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rayhan Lal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan

RESULTS

PARTICIPANT FLOW:
Period: Week 1 (First Injection)
Arm/Group | Upper Peritoneal, Then Lower Peritoneal, Then Subcutaneous | Lower Peritoneal, Then Upper Peritoneal, Then Subcutaneous
Started | 10 | 6
Received Injection | 10 | 6
Received Disallowed Medication Prior to Injection | 0 | 1
Suspension of Basal Insulin > 2 Hours Prior to Injection | 1 | 1
Achieved Induced Hypoglycemia | 4 | 4
Completed | 10 | 5
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Week 2 (Second Injection)
Arm/Group | Upper Peritoneal, Then Lower Peritoneal, Then Subcutaneous | Lower Peritoneal, Then Upper Peritoneal, Then Subcutaneous
Started | 10 | 5
Suspension of Basal Insulin > 2 Hours Prior to Injection | 1 | 1
Achieved Induced Hypoglycemia | 7 | 4
Completed | 10 | 5
Not Completed | 0 | 0
Period: Week 3 (Third Injection)
Arm/Group | Upper Peritoneal, Then Lower Peritoneal, Then Subcutaneous | Lower Peritoneal, Then Upper Peritoneal, Then Subcutaneous
Started | 10 | 5
Suspension of Basal Insulin > 2 Hours Prior to Injection | 1 | 1
Achieved Induced Hypoglycemia | 9 | 4
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Upper Peritoneal, Then Lower Peritoneal, Then Subcutaneous | Lower Peritoneal, Then Upper Peritoneal, Then Subcutaneous | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (7.1) | 38.8 (11.7) | 38.9 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 10 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 5 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Glucagon Response to Induced Hypoglycemia
Description: For each injection site we will assess the peak concentration of glucagon at time of the first induced hypoglycemic nadir.
  Analysis includes reporting groups for each type of injection, and upper and lower peritoneal injections combined (Injection- All Peritoneal).
  Participants must have achieved induced hypoglycemia to be evaluable for the primary outcome.
Time Frame: Peritoneal: Every 5 minutes for 180 minutes max; Subcutaneous: Every 15 minutes for 360 minutes max
Population: Participants with successfully induced hypoglycemia at the respective study visit
Measure: Median (Inter-Quartile Range); unit: pg/mL
Units Other Than Participants: Injections
Groups:
- Upper Peritoneal Injection: Ultra-fast acting insulin injected into the upper peritoneum
- Lower Peritoneal Injection: Ultra-fast acting insulin injected into the lower peritoneum
- Injection- All Peritoneal: Ultra-fast acting insulin injected into the peritoneum
- Subcutaneous Injection: Ultra-fast acting insulin injected subcutaneously
Arm/Group | Upper Peritoneal Injection | Lower Peritoneal Injection | Injection- All Peritoneal | Subcutaneous Injection
Number analyzed (Participants) | 8 | 11 | 13 | 13
Number analyzed (Injections) | 8 | 11 | 19 | 13
pg/mL | 4.8 [2.7 to 8.2] | 8.8 [3.4 to 12.8] | 5.8 [3.0 to 9.1] | 4.2 [2.3 to 6.3]

2. Secondary Outcome: Insulin Maximum Concentration in Plasma
Description: We will assess the maximum concentration of circulating insulin for each injection site after a median injection of 40% of each participant's total daily dose (approximately 0.25 units per kilogram of body weight).
  Analysis includes reporting groups for each type of injection, and upper and lower peritoneal injections combined (Injection- All Peritoneal).
Time Frame: Peritoneal: Every 5 minutes for 180 minutes max; Subcutaneous: Every 15 minutes for 360 minutes max
Population: Participants were excluded if they took a disallowed medication, or if the suspension of basal insulin prior to injection exceeded 2 hours.
Measure: Median (Inter-Quartile Range); unit: mU/L
Units Other Than Participants: Injections
Arm/Group | Upper Peritoneal Injection | Lower Peritoneal Injection | Injection- All Peritoneal | Subcutaneous Injection
Number analyzed (Participants) | 13 | 13 | 13 | 13
Number analyzed (Injections) | 13 | 13 | 26 | 13
mU/L | 56.81 [46.40 to 63.49] | 63.26 [37.60 to 78.84] | 56.95 [44.01 to 77.57] | 57.47 [46.84 to 69.53]

3. Secondary Outcome: Hypoglycemic Treatments Required as a Measure of Glucose Values
Description: We will compare the number of rescue treatments (2.5ml/kg 10% Dextrose) required to treat hypoglycemia <50mg/dl for each injection location of approximately 0.25u/kg ultra-rapid insulin.
  Analysis includes reporting groups for each type of injection, and upper and lower peritoneal injections combined (Injection- All Peritoneal).
Time Frame: Peritoneal: Every 5 minutes for 180 minutes max; Subcutaneous: Every 15 minutes for 360 minutes max
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Treatments
Units Other Than Participants: Injections
Groups:
- Peritoneal Injection: Ultra-fast acting insulin injected into the peritoneum
Arm/Group | Upper Peritoneal Injection | Lower Peritoneal Injection | Peritoneal Injection | Subcutaneous Injection
Number analyzed (Participants) | 13 | 13 | 13 | 13
Number analyzed (Injections) | 13 | 13 | 26 | 13
Treatments | 1 [0 to 2] | 1 [1 to 1] | 1 [0 to 1] | 3 [3 to 4]

4. Secondary Outcome: Time Until Maximum Insulin Concentration in Plasma
Description: We will assess time until the maximum concentration of circulating insulin for each injection site after a median injection of 40% of each participant's total daily dose (approximately 0.25 units per kilogram of body weight).
  Analysis includes reporting groups for each type of injection, and upper and lower peritoneal injections combined (Injection- All Peritoneal).
Time Frame: Peritoneal: Every 5 minutes for 180 minutes max; Subcutaneous: Every 15 minutes for 360 minutes max
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: minutes
Units Other Than Participants: Injections
Arm/Group | Upper Peritoneal Injection | Lower Peritoneal Injection | Injection- All Peritoneal | Subcutaneous Injection
Number analyzed (Participants) | 13 | 13 | 13 | 13
Number analyzed (Injections) | 13 | 13 | 26 | 13
minutes | 35 [25 to 40] | 25 [20 to 40] | 30 [20 to 40] | 60 [45 to 75]

ADVERSE EVENTS:
Time Frame: Average approximately 2 months (may have been up to 13 months).
Arm/Group | Upper Peritoneal Injection | Lower Peritoneal Injection | Subcutaneous Injection
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT04416737/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT04416737/ICF_000.pdf